CLINICAL TRIAL: NCT00692822
Title: Antimicrobial Susceptibility Patterns of Neisseria Gonorrhea Isolates in an Era of Quinolone Resistance
Brief Title: Antimicrobial Susceptibility Patterns of N. Gonorrhea Isolates in an Era of Quinolone Resistance
Status: Completed | Type: Observational
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Other Study IDs: H08011
Record Dates: First submitted 2008-06-04; First posted 2008-06-06 (Estimated); Last update posted 2012-03-07 (Estimated); Status verified 2009-02

CONDITIONS: Gonorrhea
Keywords: Neisseria gonorrheae; Antimicrobial Susceptibility; Quinolone Resistance; Sexually transmitted diseases
MeSH Terms: conditions — Gonorrhea; Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urethral discharge for Neisseria gonorrheae culture
Oversight: Data Monitoring Committee: No

SUMMARY:
To perform a laboratory sensitivity testing survey of antibiotic agents against Neisseria gonorrhea isolates from men with symptomatic urethritis seen at an STD clinic.

DETAILED DESCRIPTION:
Until recently, the fluoroquinolones (ofloxacin, ciprofloxacin, levofloxacin) have been the first line oral agents for the empiric treatment of gonorrhea. The prevalence of quinolone resistant Neisseria gonorrheae (QRNG) has been rising since 2000. In 2006, the CDC updated its guidelines to include recommendations against the use of quinolones for treatment of Neisseria gonorrheae. Ceftriaxone (available only by intravenous or intramuscular route) was named as the first line treatment for urogenital and pharyngeal disease. Availability, in the United States, of the other two CDC recommended agents cefixime (oral) and spectinomycin (IM) has been nonexistent.

At this time, there is little data on the in-vitro (laboratory test) susceptibility of antibiotics against gonorrhea, particularly oral drugs. The purpose of this study is to collect specimens of gonorrhea in a non-invasive swab manner from men with symptomatic urethral discharges for laboratory sensitivity testing against a wide array of antibiotic agents.

Specific Aims:

To perform a laboratory sensitivity testing survey of antibiotic agents against Neisseria gonorrhea isolates from men with symptomatic urethritis seen at a Duval County STD clinic .

ELIGIBILITY:
Inclusion Criteria:

* Men between the ages of 18 to 80 years old with suspected urethral gonorrhea by symptoms or gram stained smear

Exclusion Criteria:

* Patients less than 18 years old or greater than 80 years old
* Inability to give an informed consent

Ages: 18 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male patients seen in the Duval County Sexually Transmitted Diseases Clinic with smears positive for gram negative diplococci or unexplained pyuria
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2008-06; Primary Completion 2010-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christina L Bailey, MD, Principal Investigator — University of Florida; Nilmarie Guzman, MD, Principal Investigator — University of Florida
Locations (1):
- Boulevard Comprehensive Care Center, Jacksonville, Florida, United States

REFERENCES:
- [Background] Weinstock H, Berman S, Cates W Jr. Sexually transmitted diseases among American youth: incidence and prevalence estimates, 2000. Perspect Sex Reprod Health. 2004 Jan-Feb;36(1):6-10. doi: 10.1363/psrh.36.6.04. PMID 14982671
- [Background] Newman LM, Moran JS, Workowski KA. Update on the management of gonorrhea in adults in the United States. Clin Infect Dis. 2007 Apr 1;44 Suppl 3:S84-101. doi: 10.1086/511422. PMID 17342672
- [Background] Tapsall JW, Shultz TR, Limnios EA, Donovan B, Lum G, Mulhall BP. Failure of azithromycin therapy in gonorrhea and discorrelation with laboratory test parameters. Sex Transm Dis. 1998 Nov;25(10):505-8. doi: 10.1097/00007435-199811000-00002. PMID 9858344
- [Background] Ito M, Yasuda M, Yokoi S, Ito S, Takahashi Y, Ishihara S, Maeda S, Deguchi T. Remarkable increase in central Japan in 2001-2002 of Neisseria gonorrhoeae isolates with decreased susceptibility to penicillin, tetracycline, oral cephalosporins, and fluoroquinolones. Antimicrob Agents Chemother. 2004 Aug;48(8):3185-7. doi: 10.1128/AAC.48.8.3185-3187.2004. PMID 15273147
- [Background] Centers for Disease Control and Prevention. Sexually Transmitted Disease Surveillance, 2004. Atlanta, GA: US Dept of Health ands Human Services, September 2005
- [Background] Hook EW III, Handsfield HH. Gonococcal infections in the adult. In: Holmes KK, Sparling PF, Mardh P, et al. Sexually Transmitted Diseases . 3rd ed. New York: Mc Graw Hill, 1999: 451-66
- [Background] Chin J. Control of Communicable Diseases Manual. 17th ed. American Public Health Association, 2000:223-228
- [Background] Sexually transmitted diseases treatment guidelines 2002. Centers for Disease Control and Prevention. MMWR Recomm Rep. 2002 May 10;51(RR-6):1-78. PMID 12184549